CLINICAL TRIAL: NCT02804412
Title: Constraint Induced Aphasia Therapy in Stroke Patients in Acute Stage.
Brief Title: Aphasia Therapy: Factors of Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Hartwig Woldag, Head of departement NRZ Leipzig, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRZ-CIAT
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Aphasia
Keywords: communication disorders; language and speech disorder rehabilitation; stroke
MeSH Terms: conditions — Aphasia; Communication Disorders; Language; Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): Patients received a standard, house-typical aphasia therapy in single and group therapy sessions
  Interventions: Other: Control group
- CIAT-group (Experimental): Patients received constraint-induced aphasia therapy.
  Interventions: Other: CIAT-group
- communication treatment group (CTG) (Active Comparator): Patients received aphasia group therapy without constraints
  Interventions: Other: communication treatment group (CTG)

INTERVENTIONS:
Other: Control group — This is the control group with 14 h treatment over 10 workdays.
  Arms: Control group
Other: CIAT-group — Examine the efficacy of CIAT (30 h over 10 workdays) versus Control-group and communication treatment group.
  Arms: CIAT-group
Other: communication treatment group (CTG) — Examine the efficacy of CTG (30h over 10 wokrdays) versus CIAT-group and control group
  Arms: communication treatment group (CTG)

SUMMARY:
Constraint-induced aphasia therapy (CIAT) has proven effective in stroke patients. It has remained unclear, however, whether intensity of therapy or constraint is the relevant factor. This study will give an answer to this question to improve speech and language therapy.

DETAILED DESCRIPTION:
Although there is clear evidence that aphasia therapy is effective, questions remain as to the intensity of administered therapy, the preferred therapeutic approach and its initiation with regard to stroke onset. CIAT is a a high intense group therapy administered over 2 weeks. Additionally, patients have to communicate solely in spoken words or sentences (constraint). This study compares CIAT with an approach of the same intensity without constraints and a less intense house-typical therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* first ever stroke
* suffering from aphasia

Exclusion Criteria:

* severe cognitive or attentional impairments
* severe depression
* left-handedness
* severe dysarthria
* apraxia of speech
* severe deafness
* additional neurological diseases affecting speech (e.g. Parkinson's disease)

Ages: 39 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change of aphasia by Aachener Aphasia Test (AAT) | pretreatment and within 24 h post intervention

SECONDARY OUTCOMES:
Change of Communication Activity Log (CAL) | pretreatment and within 24 h post intervention
  The CAL is a two-part questionnaire rating the amount and the quality of daily communication on a six-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig Woldag, PhD, Principal Investigator — NRZ Leipzig

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woldag H, Voigt N, Bley M, Hummelsheim H. Constraint-Induced Aphasia Therapy in the Acute Stage: What Is the Key Factor for Efficacy? A Randomized Controlled Study. Neurorehabil Neural Repair. 2017 Jan;31(1):72-80. doi: 10.1177/1545968316662707. Epub 2016 Aug 9. PMID 27506677